CLINICAL TRIAL: NCT04685603
Title: Adaptive Phase I Clinical Trial of Preventive Vaccine Consisting of Autologous Dendritic Cells Previously Incubated With S-protein From SARS-CoV-2, in Subjects Negative for COVID-19 Infection and Anti-SARS-CoV-2 Antibodies
Brief Title: Dendritic Cell Vaccine to Prevent COVID-19
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia-MoH (Other Government)
Collaborators: Aivita Biomedical, Inc. (Industry); PT AIVITA Biomedika Indonesia (Unknown); National Institute of Health Research and Development, Ministry of Health Republic of Indonesia (Other); RSUP Dr. Kariadi Semarang, indonesia (Unknown); Faculty of Medicine University of Diponegoro, Indonesia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CL-COV-P02-ID; U1111-1263-0568 (Other: WHO-UTN)
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: COVID-19
Keywords: covid-19; vaccine; dendritic cell
MeSH Terms: conditions — COVID-19 | interventions — AV-COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: Autologous dendritic cells previously loaded ex vivo with SARS-CoV-2 spike protein
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- AV-COVID-19 (0.1 mg antigen, 0 mcg GMCSF) (Experimental): Autologous dendritic cells previously loaded with 0.1 mg SARS-CoV-2 spike protein, admixed with 0 mcg GM-CSF
  Interventions: Biological: AV-COVID-19
- AV-COVID-19 (0.33 mg antigen, 0 mcg GM-CSF) (Experimental): Autologous dendritic cells previously loaded with 0.33 mg SARS-CoV-2 spike protein, admixed with 0 mcg GM-CSF
  Interventions: Biological: AV-COVID-19
- AV-COVID-19 (1.0 mg antigen, 0 mcg GMCSF) (Experimental): Autologous dendritic cells previously loaded with 1.0 mg SARS-CoV-2 spike protein, admixed with 0 mcg GM-CSF
  Interventions: Biological: AV-COVID-19
- Experimental: AV-COVID-19 (0.1 mg antigen, 250 mcg GM-CSF) (Experimental): Autologous dendritic cells previously loaded with 0.1 mg SARS-CoV-2 spike protein, admixed with 250 mcg GM-CSF
  Interventions: Biological: AV-COVID-19
- AV-COVID-19 (0.33 mg antigen, 250 mcg GM-CSF) (Experimental): Autologous dendritic cells previously loaded with 0.33 mg SARS-CoV-2 spike protein, admixed with 250 mcg GM-CSF
  Interventions: Biological: AV-COVID-19
- AV-COVID-19 (1.0 mg antigen, 250 mcg GM-CSF) (Experimental): Autologous dendritic cells previously loaded with 1.0 mg SARS-CoV-2 spike protein, admixed with 250 mcg GM-CSF
  Interventions: Biological: AV-COVID-19
- AV-COVID-19 (0.1 mg antigen, 500 mcg GM-CSF) (Experimental): Autologous dendritic cells previously loaded with 0.1 mg SARS-CoV-2 spike protein, admixed with 500 mcg GM-CSF
  Interventions: Biological: AV-COVID-19
- AV-COVID-19 (0.33 mg antigen, 500 mcg GM-CSF) (Experimental): Autologous dendritic cells previously loaded with 0.33 mg SARS-CoV-2 spike protein, admixed with 500 mcg GM-CSF
  Interventions: Biological: AV-COVID-19
- AV-COVID-19 (1.0 mg antigen, 500 mcg GM-CSF) (Experimental): Autologous dendritic cells previously loaded with 1.0 mg SARS-CoV-2 spike protein, admixed with 500 mcg GM-CSF
  Interventions: Biological: AV-COVID-19

INTERVENTIONS:
Biological: AV-COVID-19 — Autologous dendritic cells previously loaded ex vivo with SARS-CoV-2 spike protein

SUMMARY:
This is an adaptive Phase I trial of a vaccine consisting of autologous dendritic cells previously loaded ex vivo with SARS-CoV-2 spike protein, with or without GM-CSF, to prevent COVID-19 in adults.

DETAILED DESCRIPTION:
Subjects eligible for treatment will be those who at baseline, are not actively infected with SARS-CoV-2, have no evidence of prior infection with SARSCoV- 2 based on serologic testing, and give informed consent for a vaccination with AV-COVID-19. The patient population will include the elderly and others at higher risk for poor outcomes after COVID-19 infection. For this reason, individuals will not be excluded solely on the basis of age, body mass index, history of hypertension, diabetes, cancer, or autoimmune disease.

After enrolling for screening, subjects will undergo a nasal swab test to exclude active COVID-19 infection and a rapid test for anti-coronavirus antibodies to exclude pre-existing anti-SARS-CoV-2 antibodies. 50 mL of blood will be collected, from which peripheral blood monocytes will be isolated and differentiated into DC before incubation with SARS-CoV-2 S-protein, during which time the protein is digested into 9 to 25 amino acid peptide sequences presented on the dendrites of DC in conjunction with histocompatibility class I and class II molecules. Safety and quality testing will be performed on a small quantity of the batch, and the remaining AV-COVID-19 will be cryopreserved for shipping to the treatment site.

Once the Study Drug is ready, if eligible, the subject will be seen at Study Week-0 for treatment. Prior to injection of the Study Drug, a nasal swab test will be collected to confirm that they are still negative for COVID-19, and blood will be drawn to determine baseline levels of anti-SARS-CoV-2 antibodies. At the treatment site, the product will be thawed and admixed with saline or (saline with GM-CSF), and within 5 hours of thawing, will be injected SC via a 25- gauge needle

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older,
2. in relatively good health with adequate physical and mental function
3. including factors associated with in increased risk for medical complications associated with COVID-19 infection or increased risk for exposure to SARS-CoV-2

Exclusion Criteria:

1. Active COVID-19 infection by PCR testing
2. Pre-existing IgG or IgM SARS-CoV-2 antibodies
3. Pregnant, Known hypersensitivity to GM-CSF
4. Known active immune deficiency disease or active HIV
5. HBV, HCV, On active treatment with corticosteroids or other immunosuppressive agent
6. Participated in previous COVID-19 vaccine study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2020-12-07 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of solicited local and systemic reactogenicity adverse events (AEs) | until follow up day 7
  Percentage of participants with solicited AEs (local, systemic) for 7 days following vaccination by severity score, duration, and peak intensity.
Safety Laboratory Values (Serum Chemistry) | until follow up day 7
  Safety laboratory values (Serum Chemistry) by FDA toxicity scoring (absolute and change from baseline where identified) at 7 days after each vaccination.
Safety Laboratory Values (Hematology) | until follow up day 7
  Safety laboratory values (Hematology) by FDA toxicity scoring (absolute and change from baseline where identified) at 7 days after each vaccination.
Frequency of any serious adverse events (SAEs) | until follow up day 365
  Percentage of participants with serious undesirable effect associated with the use of a medical product in a patient, which consist of death, life-threatening, hospitalization, disability or permanent damage, congenital anomaly/birth defect, required intervention to prevent permanent impairment or damage (devices), dan other serious important medical events
Frequency of any new-onset chronic medical conditions (NOCMCs) | until follow up day 365
  NOCMCs will be documented from the time of study vaccination through approximately 1 year after study vaccination
Frequency of medically attended adverse events (MAAEs) | until follow up day 365
  Percentage of participants with MAAEs, defined as AEs that lead to an unscheduled visit to a healthcare practitioner, through Day 365 by MedDRA classification, severity score, and relatedness.
Frequency of Unsolicited AE and Adverse Events of Special Interest (AESIs) | until follow up day 90
  Percentage of participants with unsolicited AEs (eg, treatment-emergent, serious, suspected unexpected serious, those of special interest, all MAAEs) or AESIs (potential immune-mediated medical conditions or AEs relevant to COVID-19) through the first 90 days by MedDRA classification, severity score, and relatedness.

SECONDARY OUTCOMES:
Serum IgG Antibody Levels Expressed as Geometric Mean Fold Rises (GMFRs) | until follow up day 28
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by ELISA expressed as GMFRs through Day 28.
Serum Immunoglobulin G (IgG) Antibody Levels Expressed as Geometric Mean Titers (GMTs) | until follow up day 28
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by enzyme-linked immunosorbent assay (ELISA) expressed as GMTs through Day 28.
Serum IgG Antibody Levels Expressed as Seroconversion Rates (SCRs) | until follow up day 28
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by ELISA expressed as SCRs through Day 28. SCR is the proportion of participants with ≥4-fold rises in ELISA units.
Neutralizing Antibody Activity Expressed as GMTs | until follow up day 28
  Neutralizing antibody activity as detected by microneutralization assay (MN) expressed as GMTs at multiple time points through Day 28.
Neutralizing Antibody Activity Expressed as GMFRs | until follow up day 28
  Neutralizing antibody activity as detected by MN expressed as GMFRs at multiple time points through Day 28.
Neutralizing Antibody Activity Expressed as SCRs | until follow up day 28
  Neutralizing antibody activity as detected by MN expressed as SCRs at multiple time points through Day 28.
Assessment of Cell-Mediated (T helper 1 [Th1]/T helper 2 [Th2]) Pathways | until follow up day 28
  Cell-mediated (Th1/Th2) pathways as measured by whole blood (flow cytometry) and/or in vitro peripheral blood mononuclear cell (PBMC) stimulation (eg, enzyme-linked immunospot [ELISpot], cytokine staining) with SARS-CoV-2 rS protein(s) through Day 28.
Optimal dose of SARS-CoV2 antigen and GM-CSF | until follow up month one
  Measurement of IgG in subject blood after one month
Duration of detection IgG and neutralizing antibody againts SARS-CoV-2in blood after vaccination | until follow up month 12
  Measurement of IgG and neutralizing antibody in subject blood after 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Djoko Wibisono, Dr. Internis, Principal Investigator — Rumah Sakit Pusat Angkatan Darat (RSPAD) Gatot Soebroto, Jakarta; Muhammad Karyana, Principal Investigator — National Institute of Health Research and Development
Locations (1):
- Rumah Sakit Umum Pusat Dr. Kariadi, Semarang, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No